CLINICAL TRIAL: NCT04810650
Title: A Multisectoral Strategy to Address Persistent Drivers of the HIV Epidemic in East Africa
Brief Title: SEARCH SAPPHIRE Phase A: A Multisectoral Strategy to Address Persistent Drivers of the HIV Epidemic in East Africa
Acronym: SAPPHIRE PhA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Infectious Diseases Research Collaboration, Uganda (Other); Makerere University (Other); Kenya Medical Research Institute (Other); University of California, Berkeley (Other); University College, London (Other); University of Pennsylvania (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SEARCH SAPPHIRE Phase A; U01AI150510 (NIH)
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: HIV; Hypertension; Alcohol Drinking; Maternal Child Health; Cost Effectiveness
Keywords: PrEP; PEP; HIV Treatment and Prevention; Community Health; Mobile Populations; Youth and Adolescents
MeSH Terms: conditions — Hypertension; Alcohol Drinking | interventions — Ethanol; Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel randomized trials to assess effectiveness, fidelity and cost of prevention and treatment interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- PREP/PEP at Outpatient Clinics Dynamic Prevention Intervention (Experimental)
  Interventions: Other: PrEP/PEP at Outpatient Clinics
- PREP/PEP at Outpatient Clinics Control (Active Comparator)
  Interventions: Other: Standard of Care
- PREP/PEP at Antenatal Clinics Dynamic Prevention Intervention (Experimental)
  Interventions: Other: PrEP/PEP at Antenatal Clinics
- PREP/PEP at Antenatal Clinics Control (Active Comparator)
  Interventions: Other: Standard of Care
- PREP/PEP at Community Households Dynamic Prevention Intervention (Experimental)
  Interventions: Other: PrEP/PEP at Community Households
- PREP/PEP at Community Households Control (Active Comparator)
  Interventions: Other: Standard of Care
- Mobility Dynamic Treatment Intervention (Experimental)
  Interventions: Other: Mobility Dynamic Treatment Intervention
- Mobility Control (Active Comparator)
  Interventions: Other: Standard of Care
- Healthy Living for Heavy Alcohol Users Intervention (Experimental)
  Interventions: Other: Health Living Intervention for Heavy Alcohol Users
- Heavy Alcohol Users Control (Active Comparator)
  Interventions: Other: Standard of Care
- Hypertension Linkage Intervention (Experimental)
  Interventions: Other: Hypertension Linkage
- Hypertension Linkage Control (Active Comparator)
  Interventions: Other: Standard of Care
- Hypertension Community Intervention (Experimental)
  Interventions: Other: Hypertension Community
- Hypertension Community Control (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Mobility Dynamic Treatment Intervention — 1) Access to a mobility coordinator who will assist with transfers, rescheduling, and out-of-facility refills; 2) Provision of a "travel pack" with alternative ART packaging options (e.g. ziplock bags, envelopes, pill boxes), a packing list and mobility coordinator phone contact for unplanned travel; 3) Screening at every clinic visit for planned mobility; 4) Mobile number and mobile minutes for unexpected travel; 5) Provision of longer refills (up to 6-months) for planned travel
  Arms: Mobility Dynamic Treatment Intervention
Other: Health Living Intervention for Heavy Alcohol Users — 1) Two in-person alcohol counseling sessions with support from a clinical psychologist; 2) Monthly booster phone calls
  Arms: Healthy Living for Heavy Alcohol Users Intervention
Other: Hypertension Linkage — 1) Travel voucher (financial incentive) conditional on linkage to hypertensive care; 2) Phone call reminders for missed visits
  Arms: Hypertension Linkage Intervention
Other: PrEP/PEP at Outpatient Clinics — Intervention delivered at Outpatient Clinics: Counseling and education on and choice between prevention modalities (e.g. PrEP, PEP, condoms), choice of service location, provision of a clinical officer's or nurse's mobile telephone number for immediate PEP starts any day of the week, routine assessment of barriers to initiation or adherence to PrEP/PEP, including the offer of personalized potential solutions such as choice of in-clinic or offsite service delivery, psychologic supports for traumatic experiences, and offer of concurrent, additional health or prevention related services
  Arms: PREP/PEP at Outpatient Clinics Dynamic Prevention Intervention
Other: PrEP/PEP at Antenatal Clinics — Intervention delivered at Antenatal Clinics: Counseling and education on and choice between prevention modalities (e.g. PrEP, PEP, condoms), choice of service location, provision of a clinical officer's or nurse's mobile telephone number for immediate PEP starts any day of the week, routine assessment of barriers to initiation or adherence to PrEP/PEP, including the offer of personalized potential solutions such as choice of in-clinic or offsite service delivery, psychologic supports for traumatic experiences, and offer of concurrent, additional health or prevention related services
  Arms: PREP/PEP at Antenatal Clinics Dynamic Prevention Intervention
Other: PrEP/PEP at Community Households — Intervention delivered in community by village health team: Counseling and education on and choice between prevention modalities (e.g. PrEP, PEP, condoms), choice of service location, provision of a clinical officer's or nurse's mobile telephone number for immediate PEP starts any day of the week, routine assessment of barriers to initiation or adherence to PrEP/PEP, including the offer of personalized potential solutions such as choice of in-clinic or offsite service delivery, psychologic supports for traumatic experiences, and offer of concurrent, additional health or prevention related services
  Arms: PREP/PEP at Community Households Dynamic Prevention Intervention
Other: Standard of Care — Local country standard of care protocols
  Arms: Heavy Alcohol Users Control; Hypertension Community Control; Hypertension Linkage Control; Mobility Control; PREP/PEP at Antenatal Clinics Control; PREP/PEP at Community Households Control; PREP/PEP at Outpatient Clinics Control
Other: Hypertension Community — Hypertension care delivered at home with clinician telehealth, facilitated by lay health worker to measure blood pressure and deliver medications
  Arms: Hypertension Community Intervention

SUMMARY:
The randomized trials in this record will assess effectiveness, fidelity and cost of prevention and treatment interventions for HIV and hypertension with the objective of informing a population-based study of multi-sectored, multi-disease interventions for HIV.

DETAILED DESCRIPTION:
The study will conduct randomized trials to assess effectiveness, fidelity and cost of prevention and treatment interventions. The study will conduct two randomization trials to evaluate dynamic treatment interventions tailored to the needs of heavy alcohol users and mobile populations. The study will conduct three randomized trials to evaluate dynamic choice prevention interventions delivered in the context of antenatal clinics, the outpatient department, and in the community delivered by village health teams. The trial will conduct a randomized trial to evaluate a linkage intervention for patients with hypertension and a randomized trial to evaluate a clinic vs. community based intervention for hypertension.

ELIGIBILITY:
INDIVIDUAL LEVEL INCLUSION CRITERIA FOR COMPONENT INTERVENTIONS

PrEP/PEP at Outpatient Clinics

1. Age ≥15 years
2. HIV-negative
3. Current or anticipated risk for HIV-infection

PrEP/PEP at Antenatal Clinics

1. Age ≥15 years
2. HIV-negative
3. Current or anticipated risk for HIV-infection

PrEP/PEP at Community Households

1. Age > 15 years
2. HIV-negative
3. Current or anticipated risk for HIV-infection

Mobility Dynamic Treatment Intervention

1. Age ≥15 years
2. HIV-positive
3. HIV RNA non-suppression (>400 c/mL in the prior 12 months) or missed 2 visits in past 12 months or missed 2 visits in past 12 months or no VL measured in past 12 months
4. Travel outside the community ≥2 times in past 12 months
5. Enrolled or new to care in a study clinic

Healthy Living Intervention for Heavy Alcohol Users

1. Age ≥18 years
2. HIV-positive
3. HIV RNA non-suppression (>400 c/mL in the prior 12 months) or missed clinic visits (>2 weeks or <=90 days from last scheduled clinic visit) within past 6 months, or out of care without return to care (>90 days from last scheduled clinic visit) within past 6 months
4. Heavy alcohol use per AUDIT-C tool (scores of ≥4 for men, and ≥3 for women)
5. Enrolled or new to care in a study clinic

Hypertension Linkage Intervention

1. Age ≥25 years
2. Blood pressure ≥140/90 mmHg on three repeated measurements during community-based hypertension screening
3. Resident (by self-report) within catchment area of referral health center

Community Hypertension Intervention

1. Age >=40
2. Blood pressure ≥160/100 on average of 2nd and 3rd measurements at initial screening
3. Sustained blood pressure elevation to ≥140/90 at initial clinic enrollment visit

INDIVIDUAL LEVEL EXCLUSION CRITERIA FOR COMPONENT INTERVENTIONS

PrEP/PEP at Outpatient Clinics

1. <15 years of age
2. Unable to provide consent or parental co-consent as per country guidelines
3. Participation in another Phase A RCT intervention component

PrEP/PEP at Antenatal Clinics

1. <15 years of age
2. unable to provide consent or parental co-consent as per country guidelines
3. Participation in another Phase A RCT intervention component

PrEP/PEP at Community Households

1. <15 years of age
2. unable to provide consent or parental co-consent as per country guidelines
3. Participation in another Phase A RCT intervention component

Mobility Dynamic Treatment intervention

1. <15 years of age
2. Participation in another Phase A RCT intervention component

Healthy Living Intervention for Heavy Alcohol Users

1. <18 years of age
2. Participation in another Phase A RCT intervention component
3. No access to mobile phone

Hypertension Linkage Intervention

1. <25 years of age
2. Plan to out-migrate from the catchment area of referral health center within 30 days of screening visit
3. Already engaged in hypertensive care (by self-report)
4. Blood pressure measure of ≥180/110 mmHg during screening symptoms of hypertensive emergency

Community Hypertension Intervention

1. Pregnancy
2. Co-morbidities that preclude home monitoring

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2233 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Principal Investigator — University of California, San Francisco; Moses Kamya, MBChB, PhD, Principal Investigator — Makerere University; Maya Petersen, PhD, Principal Investigator — University of California, Berkeley
Locations (2):
- GPRT / SEARCH Office, Kisumu, Kenya
- IDRC Southwest Uganda, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koss CA, Ayieko J, Kabami J, Balzer LB, Kakande E, Sunday H, Nyabuti M, Wafula E, Shade SB, Biira E, Opel F, Atuhaire HN, Okochi H, Ogachi S, Gandhi M, Bacon MC, Bukusi EA, Chamie G, Petersen ML, Kamya MR, Havlir DV; SEARCH study team. Dynamic choice HIV prevention intervention at outpatient departments in rural Kenya and Uganda. AIDS. 2024 Mar 1;38(3):339-349. doi: 10.1097/QAD.0000000000003763. Epub 2023 Oct 19. PMID 37861683
- [Result] Kabami J, Koss CA, Sunday H, Biira E, Nyabuti M, Balzer LB, Gupta S, Chamie G, Ayieko J, Kakande E, Bacon MC, Havlir D, Kamya MR, Petersen M; SEARCH Study Team. Randomized Trial of Dynamic Choice HIV Prevention at Antenatal and Postnatal Care Clinics in Rural Uganda and Kenya. J Acquir Immune Defic Syndr. 2024 Apr 15;95(5):447-455. doi: 10.1097/QAI.0000000000003383. Epub 2024 Mar 11. PMID 38489493
- [Result] Kakande ER, Ayieko J, Sunday H, Biira E, Nyabuti M, Agengo G, Kabami J, Aoko C, Atuhaire HN, Sang N, Owaranganise A, Litunya J, Mugoma EW, Chamie G, Peng J, Schrom J, Bacon MC, Kamya MR, Havlir DV, Petersen ML, Balzer LB; SEARCH Study Team. A community-based dynamic choice model for HIV prevention improves PrEP and PEP coverage in rural Uganda and Kenya: a cluster randomized trial. J Int AIDS Soc. 2023 Dec;26(12):e26195. doi: 10.1002/jia2.26195. PMID 38054535
- [Result] Ayieko J, Balzer LB, Inviolata C, Kakande E, Opel F, Wafula EM, Kabami J, Owaraganise A, Mwangwa F, Nakato H, Bukusi EA, Camlin CS, Charlebois ED, Bacon MC, Petersen ML, Kamya MR, Havlir DV, Chamie G; SEARCH Study Team. Randomized Trial of a "Dynamic Choice" Patient-Centered Care Intervention for Mobile Persons With HIV in East Africa. J Acquir Immune Defic Syndr. 2024 Jan 1;95(1):74-81. doi: 10.1097/QAI.0000000000003311. Epub 2023 Dec 1. PMID 38054932
- [Result] Puryear SB, Mwangwa F, Opel F, Chamie G, Balzer LB, Kabami J, Ayieko J, Owaraganise A, Kakande E, Agengo G, Bukusi E, Kabageni S, Omoding D, Bacon M, Schrom J, Woolf-King S, Petersen ML, Havlir DV, Kamya M, Hahn JA. Effect of a brief alcohol counselling intervention on HIV viral suppression and alcohol use among persons with HIV and unhealthy alcohol use in Uganda and Kenya: a randomized controlled trial. J Int AIDS Soc. 2023 Dec;26(12):e26187. doi: 10.1002/jia2.26187. PMID 38054564
- [Result] Hickey MD, Owaraganise A, Sang N, Opel FJ, Mugoma EW, Ayieko J, Kabami J, Chamie G, Kakande E, Petersen ML, Balzer LB, Kamya MR, Havlir DV. Effect of a one-time financial incentive on linkage to chronic hypertension care in Kenya and Uganda: A randomized controlled trial. PLoS One. 2022 Nov 7;17(11):e0277312. doi: 10.1371/journal.pone.0277312. eCollection 2022. PMID 36342940
- [Derived] Kabami J, Kakande E, Chamie G, Balzer LB, Petersen ML, Camlin CS, Nyabuti M, Koss CA, Bukusi EA, Kamya MR, Havlir DV, Ayieko J. Uptake of a patient-centred dynamic choice model for HIV prevention in rural Kenya and Uganda: SEARCH SAPPHIRE study. J Int AIDS Soc. 2023 Jul;26 Suppl 1(Suppl 1):e26121. doi: 10.1002/jia2.26121. PMID 37408473
- See also: SEARCH — https://www.searchendaids.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PREP/PEP at Outpatient Clinics Dynamic Prevention Intervention | PREP/PEP at Outpatient Clinics Control | PREP/PEP at Antenatal Clinics Dynamic Prevention Intervention | PREP/PEP at Antenatal Clinics Control | PREP/PEP at Community Households Dynamic Prevention Intervention | PREP/PEP at Community Households Control | Mobility Dynamic Treatment Intervention | Mobility Control | Healthy Living for Heavy Alcohol Users Intervention | Heavy Alcohol Users Control | Hypertension Linkage Intervention | Hypertension Linkage Control | Hypertension Community Intervention | Hypertension Community Control
Started | 197 | 206 | 203 | 197 | 212 | 217 | 102 | 99 | 198 (1 participant was disenrolled in error at baseline and was not included in the baseline characteristics or at risk for adverse events.) | 203 | 100 | 99 | 98 | 102
Completed | 182 | 194 | 196 | 188 | 202 | 211 | 100 | 96 | 185 | 192 | 97 (3 participants did not complete the 3-month follow-up visit but were included in the primary outcome analysis whose timeframe was 30 days.) | 99 | 93 (6 participants did not complete the Week 48 visit but were included in the primary analysis whose timeframe was 24 weeks.) | 92 (7 participants did not complete the Week 48 visit but were included in the primary analysis whose timeframe was 24 weeks.)
Not Completed | 15 | 12 | 7 | 9 | 10 | 6 | 2 | 3 | 13 | 11 | 3 | 0 | 5 | 10
Not completed — Disenrolled in error | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 1
Not completed — Moved/transferred care | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 12 | 10 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 15 | 12 | 7 | 9 | 10 | 6 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 9
Not completed — Participant declined | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PREP/PEP at Outpatient Clinics Dynamic Prevention Intervention | PREP/PEP at Outpatient Clinics Control | PREP/PEP at Antenatal Clinics Dynamic Prevention Intervention | PREP/PEP at Antenatal Clinics Control | PREP/PEP at Community Households Dynamic Prevention Intervention | PREP/PEP at Community Households Control | Mobility Dynamic Treatment Intervention | Mobility Control | Healthy Living for Heavy Alcohol Users Intervention | Heavy Alcohol Users Control | Hypertension Linkage Intervention | Hypertension Linkage Control | Hypertension Community Intervention | Hypertension Community Control | Total
Number analyzed (Participants) | 197 | 206 | 203 | 197 | 212 | 217 | 102 | 99 | 197 | 203 | 100 | 99 | 98 | 102 | 2232
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [22 to 36] | 29 [22 to 37] | 24 [20 to 29] | 24 [20 to 29] | 29 [22 to 38] | 30 [22 to 40] | 38 [31 to 42] | 36 [29 to 45] | 37 [31 to 45] | 37 [30 to 42] | 57 [47 to 69] | 56 [47 to 68] | 60 [50 to 70] | 63 [53 to 73] | 34 [25 to 45]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant enrolled in the Heavy Alcohol Use primary outcome's intervention arm was not analyzed because the individual was disenrolled in error.
  Participants
    Female | 120 | 125 | 203 | 197 | 124 | 119 | 56 | 53 | 60 | 71 | 60 | 59 | 69 | 70 | 1386
    Male | 77 | 81 | 0 | 0 | 88 | 98 | 46 | 46 | 137 | 132 | 40 | 40 | 29 | 32 | 846
Race/Ethnicity, Customized [Number; unit: Participants]
  African | 197 | 206 | 203 | 197 | 212 | 217 | 102 | 99 | 197 | 203 | 100 | 99 | 98 | 102 | 2232
Region of Enrollment [Number; unit: participants] — Population: 1 participant enrolled in the Heavy Alcohol Use primary outcome's intervention arm was not analyzed because the individual was disenrolled in error.
  participants
    Uganda | 100 | 102 | 100 | 99 | 102 | 117 | 51 | 49 | 113 | 117 | 50 | 50 | 48 | 52 | 1150
    Kenya | 97 | 104 | 103 | 98 | 110 | 100 | 51 | 50 | 84 | 86 | 50 | 49 | 50 | 50 | 1082

OUTCOME MEASURES:

1. Primary Outcome: Prevention Coverage Defined as Percentage of Follow-up Months That the Participant Used Either PrEP or PEP
Description: Primary outcome for comparison for PrEP/PEP Dynamic Prevention Intervention at outpatient clinics vs. PrEP/PEP standard of care at outpatient clinics (not applicable to other arms). Primary definition of coverage will rely on self report.
Time Frame: 48 weeks
Population: Participants who completed the Week 48 visit.
Measure: Mean (95% Confidence Interval); unit: Percentage of months
Arm/Group | PREP/PEP at Outpatient Clinics Dynamic Prevention Intervention | PREP/PEP at Outpatient Clinics Control
Number analyzed (Participants) | 182 | 194
Percentage of months | 47.5 [42.3 to 52.7] | 18.3 [14.4 to 22.1]

2. Primary Outcome: Prevention Coverage Defined as Percentage of Follow-up Months at Risk That the Participant is Protected From HIV Infection With Either PrEP or PEP
Description: Primary outcome for comparison for PrEP/PEP Dynamic Prevention Intervention at antenatal clinics vs. PrEP/PEP standard of care at antenatal clinics (not applicable to other arms). Primary definition of coverage will rely on self report.
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage of months
Arm/Group | PREP/PEP at Antenatal Clinics Dynamic Prevention Intervention | PREP/PEP at Antenatal Clinics Control
Number analyzed (Participants) | 196 | 188
Percentage of months | 70 [65 to 74] | 29 [25 to 34]

3. Primary Outcome: Prevention Coverage Defined as Proportion of Follow-up Months at Risk That the Participant is Protected From HIV Infection With Either PrEP or PEP
Description: Primary outcome for comparison for PrEP/PEP Dynamic Prevention Intervention at community households vs. PrEP/PEP standard of care at community households (not applicable to other arms). Primary definition of coverage will rely on self report.
Time Frame: 48 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage of months
Arm/Group | PREP/PEP at Community Households Dynamic Prevention Intervention | PREP/PEP at Community Households Control
Number analyzed (Participants) | 202 | 211
Percentage of months | 28.0 [23.5 to 32.4] | 0.5 [0 to 1.0]

4. Primary Outcome: Number of Participants With Viral Suppression Defined by HIV RNA<400 Cps/ml
Description: Primary outcome for comparison of Mobility Dynamic Treatment intervention vs. standard of care control (not applicable to other arms). Data collected from medical records.
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mobility Dynamic Treatment Intervention | Mobility Control
Number analyzed (Participants) | 100 | 96
Participants | 85 | 83

5. Primary Outcome: Percentage of Participants With Viral Suppression Defined by HIV RNA<400 Cps/ml
Description: Primary outcome for comparison of Healthy Living Intervention for Heavy Alcohol Users vs. standard of care control (not applicable to other arms). Data collected from medical records.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants with VL <400
Arm/Group | Healthy Living for Heavy Alcohol Users Intervention | Heavy Alcohol Users Control
Number analyzed (Participants) | 185 | 192
Percentage of participants with VL <400 | 83 [78 to 89] | 82 [77 to 87]

6. Primary Outcome: Number of Participants Who Linked to Hypertension Care
Description: Primary outcome for comparison of Hypertension linkage intervention vs. hypertension linkage control (not applicable for other arms). Linkage to hypertension care at the local government clinic within 30 days of screening positive for high blood pressure during community screening. The primary definition will rely on clinical records.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Hypertension Linkage Intervention | Hypertension Linkage Control
Number analyzed (Participants) | 100 | 99
Participants | 96 | 65

7. Primary Outcome: Percentage of Participants With Hypertension Control <140/90 mmHg
Description: Primary outcome for hypertension community treatment intervention vs. hypertension community treatment control (not applicable for other arms). Blood pressure will be measured three times using standardized procedures in all trial participants at the 24-week study visit. Hypertension is considered controlled if the average of the 2nd and 3rd measures <140 mmHg systolic and <90 mmHg diastolic.
Time Frame: 24 weeks
Population: Participants who completed the 24-week follow-up visit
Measure: Number (95% Confidence Interval); unit: Percentage of persons with HTN control
Arm/Group | Hypertension Community Intervention | Hypertension Community Control
Number analyzed (Participants) | 96 | 99
Percentage of persons with HTN control | 77 [69 to 85] | 51 [42 to 60]

ADVERSE EVENTS:
Time Frame: Between 30 days and 48 weeks depending on the primary outcome measure.
Description: Serious adverse events were reported regardless of relationship to the study intervention. Control arm participants were not contacted during the study except at baseline and at milestone visits. Other [Not Including Serious] Adverse Events were not monitored/assessed in both intervention and control arms.
Groups:
- PREP/PEP at Antenatal Clinics Dynamic Prevention Intervention: PrEP/PEP at Antenatal Clinics: Intervention delivered at Antenatal Clinics: Counseling and education on choice between prevention modalities (e.g. PrEP, PEP, condoms), choice of service location, provision of a clinical officer's or nurse's mobile telephone number for immediate PEP starts any day of the week, routine assessment of barriers to initiation or adherence to PrEP/PEP, including the offer of personalized potential solutions such as choice of in-clinic or offsite service delivery, psychologic supports for traumatic experiences, and offer of concurrent, additional health or prevention related services
Arm/Group | PREP/PEP at Outpatient Clinics Dynamic Prevention Intervention | PREP/PEP at Outpatient Clinics Control | PREP/PEP at Antenatal Clinics Dynamic Prevention Intervention | PREP/PEP at Antenatal Clinics Control | PREP/PEP at Community Households Dynamic Prevention Intervention | PREP/PEP at Community Households Control | Mobility Dynamic Treatment Intervention | Mobility Control | Healthy Living for Heavy Alcohol Users Intervention | Heavy Alcohol Users Control | Hypertension Linkage Intervention | Hypertension Linkage Control | Hypertension Community Intervention | Hypertension Community Control
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/206 | 0/203 | 0/197 | 0/212 | 0/217 | 2/102 | 2/99 | 0/197 | 1/203 | 0/100 | 0/99 | 2/98 | 1/102
Serious Adverse Events (participants affected / at risk) | 7/197 | 0/206 | 17/203 | 2/197 | 4/212 | 1/217 | 3/102 | 2/99 | 3/197 | 1/203 | 5/100 | 0/99 | 5/98 | 1/102
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PREP/PEP at Outpatient Clinics Dynamic Prevention Intervention (N=197) | PREP/PEP at Outpatient Clinics Control (N=206) | PREP/PEP at Antenatal Clinics Dynamic Prevention Intervention (N=203) | PREP/PEP at Antenatal Clinics Control (N=197) | PREP/PEP at Community Households Dynamic Prevention Intervention (N=212) | PREP/PEP at Community Households Control (N=217) | Mobility Dynamic Treatment Intervention (N=102) | Mobility Control (N=99) | Healthy Living for Heavy Alcohol Users Intervention (N=197) | Heavy Alcohol Users Control (N=203) | Hypertension Linkage Intervention (N=100) | Hypertension Linkage Control (N=99) | Hypertension Community Intervention (N=98) | Hypertension Community Control (N=102)
Death of premature infant (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Emergency caesarian section (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intimate partner violence (Social circumstances) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-term delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes Type 2 (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine fibroids (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death due to unknown illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hydatidiform mole (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spondylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incomplete abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cryptococcal meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Homicide (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Severe hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Right inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT04810650/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT04810650/SAP_001.pdf
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT04810650/ICF_002.pdf